CLINICAL TRIAL: NCT05809882
Title: High-frequency rTMS Therapy Experience
Brief Title: Study of Experience of High-frequency Repetitive Transcranial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rongjun Hospital of Hebei Province Affiliated to North China University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xinfu Wang, Principal Investigator, Rongjun Hospital of Hebei Province Affiliated to North China University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RongjunHebei001
Record Dates: First submitted 2023-03-17; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Chronic Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Experimental)
  Interventions: Device: Magstim RAPID2 neuromagnetic stimulator (Magstim) with an "8"-type coil
- the control group (Active Comparator)
  Interventions: Device: Magstim RAPID2 neuromagnetic stimulator (Magstim) with an "8"-type coil

INTERVENTIONS:
Device: Magstim RAPID2 neuromagnetic stimulator (Magstim) with an "8"-type coil — frequency range, 20 Hz; 90% motion threshold; 3 s of stimulation; a 57 s interval; 15 min of stimulation for each side, five times per week for a total of 20 times
  Arms: the study group
Device: Magstim RAPID2 neuromagnetic stimulator (Magstim) with an "8"-type coil — frequency range, 20 Hz，60% motion threshold; 3 s of stimulation; a 57 s interval; 15 min of stimulation for each side, five times per week for a total of 20 times. But with no stimulating energy output.
  Arms: the control group

SUMMARY:
Objective: To understand the personal experience of schizophrenia patients following repetitive transcranial magnetic stimulation (rTMS) and its connection with changes in mental symptoms, thereby enhancing the overall understanding of TMS.

Method: The investigators selected eligible schizophrenia patients for fixed-parameter rTMS treatment. A self-experience checklist post-TMS treatment and positive and negative symptom scales (PANSS) were applied to evaluate the treatment.

DETAILED DESCRIPTION:
The investigators recruited male subjects admitted to who met the criteria. They were divided into a control and a treatment group. A double-blind approach was adopted. The subjects were unaware of whether real/pseudo stimulation was applied, and the evaluators did not know the grouping specifics. All of the enrolled cases were tested for stimulation thresholds in the bilateral prefrontal cortex. The TMS treatment device was a Magstim RAPID2 neuromagnetic stimulator (Magstim) with an "8"-type coil. The study group was administered real stimulation. The treatment parameters were as follows: frequency range, 20 Hz; 90% motion threshold; 3 s of stimulation; a 57 s interval; 15 min of stimulation for each side, five times per week for a total of 20 times. For the control group, a 60% motion threshold was set; the remaining parameters were consistent with the study group but with no stimulating energy output. The therapeutic instrument model, appearance, operation process, and sounds when effecting treatment were the same for both groups. A self-experience checklist post-TMS treatment and positive and negative symptom scales (PANSS) were applied to evaluate the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) were aged 18-65 years;
* 2) fulfilled the diagnosis of International Classification of Diseases Edition 10 schizophrenia;
* 3) had been diagnosed with schizophrenia more than five years previously;
* 4) were in a stable condition;
* 5) whose medication remained unchanged during treatment;
* 6) who did not have a history of epilepsy (including drug-derived);
* 7) had no brain trauma or surgery history;
* 8) who accepted treatment voluntarily and provided signed informed consent for inclusion in the study

Exclusion Criteria:

* 1) showed contraindications to rTMS intervention;
* 2) had other neuropsychiatric disorders;
* 3) received non-convulsive electroshock treatment a month preceding the start of the study;
* 4) indicated an impulse for attacking actions and engaged in destructive and self-harming behavior;
* 5) experienced generalized or electricity-related delusionsof reference,influence, andpersecution.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Self-experience checklist post- transcranial magnetic stimulation treatment | Half an hour
  Self-experience checklist post- transcranial magnetic stimulation treatment: In the present study, "self-experience" refers to an evaluation of the changes in a patient's self-perception before and after TMS treatment.
positive and negative symptom scales (PANSS) | Half an hour
  It included 30 entries, among which seven were positive, seven were negative, and the remaining 16 entries were general psychopathology scales for assessing the overall severity of schizophrenia using a 7-level score.
The repeatable battery for the assessment of neuropsychological status | Half an hour
  The RBANS scale included 12 test items that were summarized into five sets of neuromental states (five factors), i.e., immediate memory (vocabulary learning and story review), visuospatial structure (graphic depiction and line positioning), language (picture-naming and semantic fluency), attention (digital breadth and symbolic numbers), and delayed memory (vocabulary recall, vocabulary ecognition, story recall, and graphic recall).
The Insight and Treatment Attitudes Questionnaire (ITAQ) | Half an hour
  it includes the subject's understanding of the disease and their attitude towards treatment. A higher score indicated that a patient had better self-knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Rongjun Hospital of Hebei Province Affiliated to North China University of Science and Technology, Baoding, Hebei, China